CLINICAL TRIAL: NCT00984412
Title: Allo-allo Tandem Matched Stem Cell Transplantation (AATT) for the Treatment of Patients With Refractory Acute Leukemia; a Feasibility Phase I/II Study
Brief Title: Allo-Allo Tandem Bone Marrow Transplant (BMT)
Acronym: AATT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, SHAPIRA MICHAEL, Prof shapira, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MYS-07-HMO-CTIL
Record Dates: First submitted 2009-09-06; First posted 2009-09-25 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Refractory Acute Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AATT (Experimental)
  Interventions: Procedure: Allogeneic hematopoietic stem-cell-transplantation

INTERVENTIONS:
Procedure: Allogeneic hematopoietic stem-cell-transplantation — 2 allogeneic BMTs 6 weeks apart

SUMMARY:
Refractory acute leukemia (AL) occurs in a significant percentage of the AL patients and presents a therapeutic challenge. Allogeneic stem cell transplantation (allo-SCT) is the only curative option for these patients. Although many of the patients with refractory AL that undergo myeloablative SCT initially achieve complete remission, most relapse later on, and the long-term disease free survival is poor. In order to achieve better leukemic control, most transplant centers employ post transplant early withdrawal of the anti-GVHD immunosuppression; hence exposing the patients to high risk of GVHD associated morbidity and mortality. This study will try to address this common scenario, namely early and late relapse. The investigators will try to attain better leukemic control by re-inducing the patients, 6 weeks after the 1st transplant with further myeloablative treatment (busulfex and thiotepa) followed by allogeneic stem cell support (transplant II).

DETAILED DESCRIPTION:
The effects of feasibility oExperimental design and methods f allo-allo tandem matched stem cell transplantation (AATT) in patients with refractory leukemia will be evaluated in a clinical setting. The current study is limited only for patients with refractory disease that received and failed up to 2 lines of salvage therapy, in good performance status and younger than 50 years old. Only patients that will achieve complete remission after transplant I, will have no major organ dysfunction and with acceptable performance status, will be treated with transplant II. Close monitoring with strict stopping rules including in case of excess transplant related morality, acute or chronic GVHD or graft failure will be employed.

Treatment schedule:

15 patients (divided into 2 cohorts, see below) with matched family member or unrelated donor will be included in single arm open phase I/II trial.

Conditioning protocol:

All patients will be prepared by the same sequential conditioning protocols:

Transplant I: Cy-TBI followed by Transplant II: Busulfan-thiotepa.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age 3-50 years old with refractory acute leukemia (primary refractory or refractory relapse I or II) unresponsive to up to 2 salvage lines with a matched donor (related or unrelated, matched defined as 8/8 HLA matching).
2. A donor willing and capable of donating peripheral blood stem cells and preferably also bone marrow cells, and lymphocytes if indicated.
3. Each patient / patient's guardian must sign written informed consent.
4. Patients must have an ECOG PS ≤ 1; Creatinine <1.5 mg/dl; Ejection fraction >45%; DLCO >70% of predicted; Serum bilirubin <2 mg/dl; elevated GPT or GOT < 2 x normal values before transplant I.

Exclusion Criteria:

1. Not fulfilling any of the inclusion criteria.
2. In complete or very good partial remission.
3. Beyond 2nd relapse.
4. Received > 2 lines of salvage therapy.
5. Active CNS involvement of the leukemia
6. Active life-threatening infection.
7. Overt untreated infection.
8. HIV seropositivity, Hepatitis B or C antigen positivity with evidence of active hepatitis.
9. Donor contraindication (HIV seropositive confirmed by Western Blot, Hepatitis B antigenemia, HCV, evidence of bone marrow disease, unable to donate bone marrow or peripheral blood due to concurrent medical condition).
10. Previous autologous or allogeneic stem cell transplantation.
11. Inability to comply with study requirements.

Ages: 3 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2009-11; Primary Completion 2020-04 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Transplant-related mortality (TRM) of SCT II. | 240d
Transplant-related toxicity (TRT) of SCT II. | 240d

SECONDARY OUTCOMES:
Day of neutrophil engraftment at SCT II | 240d
Day of platelet engraftment >20x109/L at SCT II | 240d
Day of platelet engraftment >50x109/L at SCT II | 240d
Acute GVHD occurrence ≥ 2 following SCT II | 100d
Time to acute GVHD following SCT II | 100d
GVHD grade following SCT II | 240d
Overall survival at 180 days from SCT II | 180d
Disease free survival at 180 days SCT II | 180d
Infections incidence | 240d
Immune reconstitution | 240d

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Derived] Tournilhac O, Altmann B, Friedrichs B, Bouabdallah K, Leclerc M, Cartron G, Turlure P, Reimer P, Wagner-Drouet E, Sanhes L, Houot R, Roussel M, Kroschinsky F, Dreger P, Viardot A, de Leval L, Rosenwald A, Gaulard P, Wulf G, Villate A, Latiere C, Elmaagacli A, Glass B, Poeschel V, Damaj G, Sibon D, Durot E, Bilger K, Banos A, Haenel M, Dreyling M, Keller U, Tiab M, Drenou B, Cornillon J, Nguyen S, Robin M, Nickelsen M, Trumper L, Lenz G, Ziepert M, Schmitz N; French Lymphoma Study Association (LYSA), the Societe Francophone de greffe de moelle et Therapie Cellulaire (SFGM-TC), and the German Lymphoma Alliance (GLA). Long-Term Follow-Up of the Prospective Randomized AATT Study (Autologous or Allogeneic Transplantation in Patients With Peripheral T-Cell Lymphoma). J Clin Oncol. 2024 Nov 10;42(32):3788-3794. doi: 10.1200/JCO.24.00554. Epub 2024 Sep 13. PMID 39270145
- [Derived] Schmitz N, Truemper L, Bouabdallah K, Ziepert M, Leclerc M, Cartron G, Jaccard A, Reimer P, Wagner E, Wilhelm M, Sanhes L, Lamy T, de Leval L, Rosenwald A, Roussel M, Kroschinsky F, Lindemann W, Dreger P, Viardot A, Milpied N, Gisselbrecht C, Wulf G, Gyan E, Gaulard P, Bay JO, Glass B, Poeschel V, Damaj G, Sibon D, Delmer A, Bilger K, Banos A, Haenel M, Dreyling M, Metzner B, Keller U, Braulke F, Friedrichs B, Nickelsen M, Altmann B, Tournilhac O. A randomized phase 3 trial of autologous vs allogeneic transplantation as part of first-line therapy in poor-risk peripheral T-NHL. Blood. 2021 May 13;137(19):2646-2656. doi: 10.1182/blood.2020008825. PMID 33512419